CLINICAL TRIAL: NCT04017546
Title: A Phase I Combination Study of CYC065 and Venetoclax in Patients with Relapsed or Refractory Acute Myeloid Leukemia or Myelodysplastic Syndromes
Brief Title: CYC065 CDK Inhibitor and Venetoclax Study in Relapsed/Refractory AML or MDS
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: Cyclacel Pharmaceuticals, Inc. (Industry)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: CYC065-03
Record Dates: First submitted 2019-07-08; First posted 2019-07-12 (Actual); Last update posted 2024-09-19 (Actual); Status verified 2024-09

CONDITIONS: AML; MDS
Keywords: CYC065; CDK2/9; venetoclax; BCL-2; MCL-1; Relapsed; Refractory; acute myeloid leukemia; myelodysplastic syndromes; AML; MDS
MeSH Terms: conditions — Recurrence; Leukemia, Myeloid, Acute; Myelodysplastic Syndromes | interventions — CYC065; venetoclax

STUDY DESIGN:
Intervention Model Description: One to 6 patients will be entered at a given CYC065 dose level. Dose escalation will be 33% after at least one patient has completed the first treatment cycle without ≥ grade 2 toxicity considered by the investigator to be related to CYC065. Upon the first occurrence of grade 2 toxicity related to CYC065, at least 3 patients will be entered at each dose level. If no DLT is observed in any patients, dose escalation will continue to be 33%. If one of 3 patients experienced a DLT at a given dose level, dose escalation will continue at 25% until MTD is reached. If 2 or more patients experienced a DLT at a given dose level, dose escalation will be stopped. At least 6 patients will be treated at MTD.
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: Yes | FDA-regulated Device: No | US Export: No

ARMS (1):
- CYC065 and venetoclax (Experimental): CYC065 will be administered intravenously via 4-hour infusion on Day 1 and Day 15. Venetoclax will be taken daily on Day 1 through Day 15. One cycle will be 28 days or 4 weeks.
  Interventions: Drug: CYC065; Drug: Venetoclax

INTERVENTIONS:
Drug: CYC065 — intravenous infusion
Drug: Venetoclax — oral capsule

SUMMARY:
A Phase I Combination Study of CYC065 and Venetoclax for Relapsed or Refractory AML or MDS

DETAILED DESCRIPTION:
This is an open-label, single arm, dose escalation study in patients with relapsed or refractory AML or MDS. Treatment will be administered on an outpatient basis and all patients will receive CYC065 over 4-hour infusion once every 2 weeks on Day 1 and Day 15 in combination with venetoclax. One treatment cycle is 4 weeks.

ELIGIBILITY:
Inclusion Criteria:

* Previously treated AML or MDS based on WHO classification and having at least 10% blasts in peripheral blood
* ECOG 0-2
* Adequate renal function
* Adequate liver function
* INR <=1.2 in patients not receiving chronic anticoagulation
* At least 2 weeks from prior cytotoxic chemotherapy, radiation therapy, major surgery or other investigational cancer therapy
* Agree to practice effective contraception

Exclusion Criteria:

* AML is of the subtype of APL or extramedullary myeloid tumor without bone marrow involvment
* Known AML involvement in CNS that is symptomatic and active
* Currently receiving radiotherapy, biological therapy, or any other investigational agents
* Uncontrolled intercurrent illness
* Pregnant or lactating
* Known to be HIV-positive
* Known active hepatitis B and/or hepatitis C infection

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 14 (Actual)
Dates: Start 2019-08-02 (Actual); Primary Completion 2022-11-15 (Actual); Study Completion 2023-04-05 (Actual)

PRIMARY OUTCOMES:
Maximum tolerated dose (MTD) | At the end of cycle 1 (each cycle is 28 days)
  Number of patients who experience dose-limiting toxicity (DLT)

SECONDARY OUTCOMES:
Pharmacokinetic effect | At the end of cycle 1 (each cycle is 28 days)
  plasma drug level
Pharmacodynamic effect | At the end of cycle 1 (each cycle is 28 days)
  MCL-1 level in peripheral white blood cells

OTHER OUTCOMES:
Anti-tumor activity | from the date of first dose of CYC065 to 4 weeks after the last dose of CYC065
  Number of patients achieving complete remission, partial remission, hematological improvement as evaluated using International Working Group (IWG) response criteria

CONTACTS AND LOCATIONS:
Overall Officials: Gautam Borthakur, MD, Principal Investigator — M.D. Anderson Cancer Center
Locations (1):
- MD Anderson Cancer Center, Houston, Texas, United States

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Derived] Frame S, Saladino C, MacKay C, Atrash B, Sheldrake P, McDonald E, Clarke PA, Workman P, Blake D, Zheleva D. Fadraciclib (CYC065), a novel CDK inhibitor, targets key pro-survival and oncogenic pathways in cancer. PLoS One. 2020 Jul 9;15(7):e0234103. doi: 10.1371/journal.pone.0234103. eCollection 2020. PMID 32645016